CLINICAL TRIAL: NCT07089472
Title: Dry Needling Versus Cyriax Technique on Pain, Paraesthesia and Functional Disability in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Faisal Javaid, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/504/08/24
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Meralgia Paresthetica; Chronic Low-back Pain (cLBP)
Keywords: Chronic low back pain; Cyriax technique; Dry needling; Functional disability; Meralgia paresthetica; Neuropathic pain; Paraesthesia; Physiotherapy
MeSH Terms: conditions — Femoral Neuropathy; Neuralgia; Paresthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): Participants in this group will receive dry needling therapy targeting muscles along the route of the lateral femoral cutaneous nerve (LFCN), including the piriformis, iliacus, tensor fascia latae, vastus lateralis, and sartorius. Each session will involve needle insertion (90 sec-2 mins) with retention for 15 minutes. Sessions will be conducted twice a week for 8 weeks (total 16 sessions). Standard physiotherapy (hot pack, EMS, stretching) will be provided alongside.
  Interventions: Behavioral: Dry Needling Therapy
- Cyriax Technique Group (Active Comparator): Participants in this group will receive the Cyriax technique (deep transverse friction massage and nerve mobilization) applied along the LFCN pathway near the anterior superior iliac spine (ASIS). Each session will involve 3-5 repetitions of mobilization, with 10-15 second holds. Sessions will be conducted twice a week for 8 weeks (total 16 sessions). Standard physiotherapy (hot pack, EMS, stretching) will be provided alongside.
  Interventions: Behavioral: Cyriax Technique

INTERVENTIONS:
Behavioral: Dry Needling Therapy — Dry needling will be applied along the lateral femoral cutaneous nerve (LFCN) pathway, targeting muscles such as piriformis, iliacus, tensor fascia latae, vastus lateralis, and sartorius. Sterile solid filiform needles (0.25x30mm and 0.30x50mm) will be inserted for 90 seconds to 2 minutes using a cone technique and retained in situ for 15 minutes. Sessions will occur twice weekly for 8 weeks, with standard physiotherapy (hot pack, EMS, and guided stretches) administered alongside.
  Arms: Dry Needling Group
Behavioral: Cyriax Technique — The Cyriax technique involves deep friction massage and mobilization of the lateral femoral cutaneous nerve (LFCN) near the anterior superior iliac spine (ASIS). Using the "pinch and roll" and deep pressure technique, therapists will apply sustained pressure along the nerve path in 3-5 repetitions per session, holding each for 10-15 seconds. Sessions will occur twice weekly for 8 weeks, alongside standard physiotherapy modalities and exercises.
  Arms: Cyriax Technique Group

SUMMARY:
This study is designed to compare the effectiveness of two physiotherapy techniques-Dry Needling and the Cyriax Technique-in people suffering from chronic low back pain (CLBP) that radiates to the outer thigh, a condition commonly known as meralgia paresthetica.

Meralgia paresthetica occurs when a nerve called the lateral femoral cutaneous nerve (LFCN) gets compressed, leading to pain, numbness, tingling, or burning sensations in the front or side of the thigh. Many patients also experience difficulty in performing daily activities because of these symptoms.

Dry Needling is a modern treatment where fine, sterile needles are inserted into specific muscles to relieve tension and improve nerve function. It is believed to release natural pain-relieving chemicals and reduce inflammation.

On the other hand, the Cyriax Technique is a manual therapy approach involving deep friction massage and gentle mobilizations targeted at the affected nerve area to reduce pressure and pain.

In this study, 80 participants between the ages of 30 and 50 years, who have had low back pain for more than three months and symptoms of nerve entrapment in the thigh, will be randomly divided into two groups. One group will receive Dry Needling therapy, and the other will receive Cyriax treatment. Both groups will also receive standard physiotherapy, including heat therapy, muscle stimulation, and stretching exercises. Treatment will continue for 8 weeks (2 sessions per week).

The aim is to evaluate and compare changes in pain, tingling/numbness (paraesthesia), and daily life functioning using recognized clinical tools such as the Visual Analogue Scale (VAS), Neuropathic Pain Symptom Inventory (NPSI), and the Roland-Morris Disability Questionnaire (RMDQ). Data will be collected at the beginning, and then again after 2, 4, and 8 weeks.

This research will help determine which therapy-Dry Needling or Cyriax-is more effective in treating patients with this type of nerve-related back and thigh pain. The findings may guide physiotherapists and healthcare providers in choosing the most suitable treatment for managing meralgia paresthetica in chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) with radiating symptoms to the anterolateral thigh, often due to meralgia paresthetica (MP), represents a complex clinical presentation with both musculoskeletal and neuropathic components. MP results from entrapment or irritation of the lateral femoral cutaneous nerve (LFCN), leading to symptoms such as numbness, tingling, burning sensations, and pain in the outer thigh. These symptoms can significantly impair quality of life and physical functioning.

This randomized controlled trial aims to compare two physiotherapeutic interventions-Dry Needling (DN) and the Cyriax Technique-with respect to their impact on pain relief, reduction of paraesthesia, and improvement in functional disability among patients with MP secondary to CLBP.

Participants will be screened based on strict inclusion and exclusion criteria. Eligible participants will be adults aged 30-50 years, diagnosed with CLBP lasting more than three months and exhibiting characteristic symptoms of MP. Exclusion criteria include prior spinal surgery, coagulopathies, serious neurological disorders, or contraindications to dry needling.

After obtaining informed consent, participants will be randomly allocated to either the experimental group (DN) or control group (Cyriax) using computer-generated randomization. Both groups will receive 16 treatment sessions over 8 weeks (2 sessions per week), in addition to standard physiotherapy consisting of heat therapy, electrical muscle stimulation, and targeted exercises.

The dry needling group will receive intramuscular stimulation along the anatomical route of the LFCN, targeting muscles including piriformis, psoas major, iliacus, tensor fasciae latae, vastus lateralis, and sartorius. Aseptic technique using solid filiform needles will be followed, with each needle retained in situ for 15 minutes per session.

The Cyriax group will receive deep transverse friction massage along the LFCN pathway, focused around the anterior superior iliac spine (ASIS), with repeated mobilizations aimed at releasing nerve entrapment and relieving local tissue tension.

Blinding will be maintained at the assessor level to reduce bias. Outcomes will be evaluated using standardized tools:

Visual Analogue Scale (VAS) for pain intensity,

Neuropathic Pain Symptom Inventory (NPSI) for paraesthesia,

Roland-Morris Disability Questionnaire (RMDQ) for functional disability.

These assessments will be conducted at baseline, 2nd, 4th, and 8th weeks of the intervention period. The study is powered at 80% with a 95% confidence interval to detect statistically significant between-group differences. Statistical analysis will be performed using SPSS, with ANOVA applied for both intra- and inter-group comparisons.

This trial is expected to provide clinically meaningful insights into which physiotherapy technique yields better therapeutic outcomes in MP associated with chronic low back pain. It will also contribute to evidence-based practice by addressing a gap in the comparative literature for these two commonly used interventions in musculoskeletal and peripheral nerve-related pain management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic low back pain (time to onset ≥ 3 months) (Erbay, 2002).
* Roland Morris Disability Questionnaire score ≥ 4 (Lara-Palomo et al., 2022).
* CLBP radiating to Anterolateral thigh with symptoms of numbness tingling (de Ruiter et al., 2023).

Exclusion Criteria:

* Patients with sensory and/or coagulation disorders (Lara-Palomo et al., 2022).
* A history of spinal surgery, heart complications, concurrent severe central or peripheral nervous system disease (de Ruiter et al., 2023).
* Epilepsy, needle phobia, serious pathologies that can be the main cause of chronic low back pain other than meralgia parasthetica (Lara-Palomo et al., 2022).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analogue Scale (VAS) | Baseline, 2nd week, 4th week, and 8th week
  Pain intensity will be assessed using the Visual Analogue Scale, a 10-cm line ranging from "no pain" to "worst possible pain." Participants will mark their pain level at each assessment point.
Change in Paraesthesia Measured by Neuropathic Pain Symptom Inventory (NPSI) | Baseline, 2nd week, 4th week, and 8th week
  Paraesthesia symptoms including tingling, burning, and numbness will be assessed using the NPSI, a self-report tool evaluating intensity and frequency of neuropathic pain symptoms.
Change in Functional Disability Measured by Roland-Morris Disability Questionnaire (RMDQ) | Baseline, 2nd week, 4th week, and 8th week
  Functional disability will be assessed using the RMDQ, a 24-item self-report questionnaire measuring the impact of low back pain on daily activities. Higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Ruiter GCW, Oosterhuis JWA, Vissers TFH, Kloet A. Unusual causes for meralgia paresthetica: systematic review of the literature and single center experience. Neurosurg Rev. 2023 May 6;46(1):107. doi: 10.1007/s10143-023-02023-2. PMID 37148363